CLINICAL TRIAL: NCT04391842
Title: Sustained Acoustic Medicine (SAM) Combined With a Diclofenac Ultrasound Coupling Patch for Knee Osteoarthritis
Acronym: SAM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HF-01
Record Dates: First submitted 2020-02-17; First posted 2020-05-18 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Osteo Arthritis Knee; Arthritis
Keywords: low-intensity ultrasound; drug delivery; sonophoresis; transdermal drug delivery; Non-Steroidal anti-inflammatory Drugs; sustained acoustic medication; low intensity continuous ultrasound
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental: SAM ultrasound and diclofenac patch (Experimental): Patients receive treatment from the SAM Ultrasonic Diathermy Device for 4 hours every day for 7 days combined with 1% diclofenac patch. The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Combination Product: Sustained Acoustic Device with 1% Diclofenac patch

INTERVENTIONS:
Combination Product: Sustained Acoustic Device with 1% Diclofenac patch — Patients apply the Sam Ultrasonic Diathermy Device daily for 4 hours of continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2 with 1% diclofenac patch
  Other Names:
  * ZetrOZ ultrasound device
  * wearable ultrasound device
  * long duration ultrasound
  * LITUS device
  * long duration low intensity device

SUMMARY:
The purpose of this study is to measure the effectiveness of Sustained Acoustic Medicine (SAM) treatment combined with diclofenac ultrasound coupling gel in patients with stage II and stage III knee osteoarthritis. The ability of the device to reduce pain, increase mobility, increase function of the affected leg, and improve quality of life in patients with knee osteoarthritis will be evaluated.

DETAILED DESCRIPTION:
This is a seven day study to clinically evaluate the effectiveness of the Sustained Acoustic Medicine (SAM) device combined with diclofenac on symptoms of patients suffering from knee osteoarthritis. The class-II device, sam® has been FDA-cleared for home use. On the first day of the study, baseline data will be collected as patients report pain score before treatment. During the following 6 days, patients will self-apply the wearable SAM device with diclofenac patch to their affected knee for 4 hours daily. Each day of the study, pain scores will be recorded immediately before application of SAM device as well as 30 minutes, 2-hours and 4-hours after applying the device. A quality of life and function assessment will be performed prior to the patient beginning the protocol and at the conclusion of the protocol.

Up to 32 subjects will be recruited from neighboring communities to the study sites. The study is designed to reach a target patient population which includes rural citizens and socioeconomic disadvantaged individuals.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed mild to moderate knee osteoarthritis (KL Grade 2-3) based on fixed-flexion x-ray radiological findings for osteophytes and joint space narrowing within the past 12 months
* Fulfill the American College of Rheumatology clinical and radiological diagnostic criteria for knee OA
* 45-85 years of age
* Report a frequent pain score between 3-7 (NRS range: 0-10) during the week preceding enrollment
* Report that knee pain negatively affects quality of life
* Willing not to use any cream, gel, or topical solution during the administration of treatment other than the approved ultrasound 1% diclofenac gel provided to the subject at the initiation of the study
* Deemed appropriate by their physician or by the study site physician to participate

Exclusion Criteria:

* Cannot successfully demonstrate the ability to put on and take off the device
* Display any condition which, in the judgment of the investigator, would make participation in the study unacceptable, including, but not limited to, the subject's ability to understand and follow instructions.
* Have severe OA or have little to no cartilage in the knee
* Have knee replacement, other surgical intervention, or hyaluronidase injection in the affected knee in the past 6 months
* Are non-ambulatory
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening
* Modify their medications during the course of the study (medications and doses must remain constant throughout the study)
* Currently taking steroids
* Have contraindication to radiograph
* Have a secondary cause of arthritis (metabolic or inflammatory)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Ortiz, DO, Study Director — Medical Pain Consultants
Locations (1):
- Cayuga Medical Center -, Dryden, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madzia A, Agrawal C, Jarit P, Petterson S, Plancher K, Ortiz R. Sustained Acoustic Medicine Combined with A Diclofenac Ultrasound Coupling Patch for the Rapid Symptomatic Relief of Knee Osteoarthritis: Multi-Site Clinical Efficacy Study. Open Orthop J. 2020;14:176-185. doi: 10.2174/1874325002014010176. Epub 2020 Dec 18. PMID 33408796
- See also: Class II Medical Device — https://www.samrecover.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: SAM Ultrasound and Diclofenac Patch: Patients receive treatment from the SAM Ultrasonic Diathermy Device for 4 hours every day for 7 days combined with 1% diclofenac patch. The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Sustained Acoustic Device with 1% Diclofenac patch: Patients apply the Sam Ultrasonic Diathermy Device daily for 4 hours of continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2 with 1% diclofenac patch
  Other Names:
  * ZetrOZ ultrasound device
  * wearable ultrasound device
  * long duration ultrasound
  * LITUS device
  * long duration low intensity device
Period: Overall Study
Arm/Group | Experimental: SAM Ultrasound and Diclofenac Patch
Started | 34
Completed | 32
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: SAM Ultrasound and Diclofenac Patch
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 53.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32
Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: Pain Units on a Scale] | 4.06 (2.39)
WOMAC [Mean (Standard Deviation); unit: Units on a Scale] | 1168 (528)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Units on a Scale (0-10) 0 Being Least, 10 Being Worst Pain From Baseline
Description: Change in the self described pain units on a scale by patient at baseline and post-treatment on the range of 0 - 10, 0 being the least pain and 10 being the worst pain.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: pain units on a scale
Arm/Group | Experimental: SAM Ultrasound and Diclofenac Patch
Number analyzed (Participants) | 32
pain units on a scale | 2.00 (2.41)
Statistical Analysis 1: Comparison: Experimental: SAM Ultrasound and Diclofenac Patch; Test type: Other; p < 0.001, ANOVA

2. Secondary Outcome: Change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Scores, Ranging From 0 Being No Difficulty to 2400 Being Extreme Difficulty, From Baseline
Description: WOMAC questionnaire will be utilized (Western Ontario and McMaster Universities Arthritis Index) at baseline and post-treatment to calculate the change in the scores. WOMAC was divided into 3 categories: pain, stiffness, function and total score. The pain category consists of five scores from 0-10, 0 is no pain 10 is worst pain possible for a range of 0 - 50 points. The stiffness category consists of two scores from 0-10, 0 is no stiffness 10 is worst stiffness possible for a range of 0 - 20 points. The function score consists of 17 scores from 0-10, 0 is normal function and 10 is severely limited function, for a range of 0 - 170 points. Categories were multiplied by 10 for analysis. Total score is the sum of pain, stiffness, and function scores (range of 0 - 2400)
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Experimental: SAM Ultrasound and Diclofenac Patch
Number analyzed (Participants) | 32
scores on a scale | -353 [-508 to -195]
Statistical Analysis 1: Comparison: Experimental: SAM Ultrasound and Diclofenac Patch; Test type: Other; p < 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Through Study Completion, an average of 7 days
Description: The risks associated with this study are minimal. There were no anticipate risk for Serious Adverse Events, risk for All-Cause Mortality or risk for Other (Not Including Serious) Adverse Events.
Arm/Group | Experimental: SAM Ultrasound and Diclofenac Patch
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04391842/Prot_SAP_000.pdf